CLINICAL TRIAL: NCT00204269
Title: Three-Year Trial on a New Testosterone Gel: Clinical Efficacy, Tolerability and Compliance
Brief Title: Three-Year Trial on a New Testosterone Gel
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRM 2002/37; TGT-04/2002
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-05-15 (Estimated); Status verified 2006-05

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Testosterone; Substitution
MeSH Terms: conditions — Hypogonadism

INTERVENTIONS:
Drug: Testosterone Gel Wolff

SUMMARY:
The objective of the study is to examine the efficacy and tolerability of a three-year-Testosterone replacement therapy in hypogonadal patients as well as the patient's compliance. The replacement therapy will be performed with a new Testosterone Gel examined in previous trials as Testosteron Gel Wolff.

DETAILED DESCRIPTION:
The objective of the study is to examine the efficacy and tolerability of a three-year-Testosterone replacement therapy in hypogonadal patients as well as the patient's compliance. The replacement therapy will be performed with a new Testosterone Gel examined in previous trials as Testosteron Gel Wolff (TGW).

A minimum of 100 patients will be recruited and evenly distributed to two treatment arms. 1st arm: dermal (non-scrotal) application of TGW. 2nd arm: scrotal application of TGW.

ELIGIBILITY:
Inclusion Criteria:

men with

* hypergonadotropic hypogonadism
* hypogonadotropic hypogonadism
* late-onset hypogonadism

combined with an initial Testosterone serum level of < 11 nmol/l

Exclusion Criteria:

* known or suspected carcinoma of the prostate
* clinically relevant abnormalities in clinical chemistry or haematology
* any severe medical conditions at the opinion of the investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-01; Study Completion 2006-09

PRIMARY OUTCOMES:
testosterone levels

SECONDARY OUTCOMES:
hormones
sexual function and mood disorder (questionnaire)
compliance (drug accountability)

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Nieschlag, Prof. Dr., Principal Investigator — Institute of Reproductive Medicine of the University
Locations (15):
- Germany (15):
  - University Clinic Charité, Division of Urology, Berlin
  - Franziskus-Hospital, Division of Urology, Bielefeld
  - University Clinic Bonn, Division of Dermatology, Bonn
  - Medical University Clinic II, Division of Internal Medicine/Andrology, Cologne
  - University Clinic Essen, Division of Internal Medicine, Essen
  - J.-W. Goethe University, Medical Clinic I, Division of Internal Medicine, Frankfurt
  - University Clinic Giessen, Division of Dermatology/Andrology, Giessen
  - University Clinic Halle Wittenberg, Division of Urology/Andrology, Halle
  - Endokrinologikum Hamburg, Hamburg
  - University Medical Clinic Hannover, Hanover
  - University Clinic Leipzig, Division of Dermatology/Andrology, Leipzig
  - Otto-von-Guerike-University, Clinic of Endocrinology, Magdeburg
  - Phillips-University-Clinic Marburg, Division of Dermatology/Andrology, Marburg
  - Insitute of Reproductive Medicine of the University, Münster
  - Private Practice of Urology, Nuremberg

REFERENCES:
- [Background] Kuhnert B, Byrne M, Simoni M, Kopcke W, Gerss J, Lemmnitz G, Nieschlag E. Testosterone substitution with a new transdermal, hydroalcoholic gel applied to scrotal or non-scrotal skin: a multicentre trial. Eur J Endocrinol. 2005 Aug;153(2):317-26. doi: 10.1530/eje.1.01964. PMID 16061839